CLINICAL TRIAL: NCT03667157
Title: Influence of Methylprednisolone Pulse Therapy on Liver Function in Patients With Graves' Orbitopathy
Brief Title: Liver Function After Intravenous Methylprednisolone Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Miskiewicz, Assistant professor, Medical University of Warsaw
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IVMPLiver
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Graves Disease; Graves Ophthalmopathy; Liver Diseases; Liver Failure; Liver Injury; Liver Dysfunction; Liver Insufficiency; Acute Liver Failure; Acute Liver Injury; Acute Liver Injury, Drug Induced; Methylprednisolone Adverse Reaction; Glucocorticoids Toxicity; Dysthyroid Orbitopathy; Dysthyroid Ophthalmopathy
Keywords: Graves Disease; Graves Ophthalmopathy; Dysthyroid Orbitopathy; Liver Failure; Liver Injury; Acute Liver Failure; Acute Liver Injury; Methylprednisolone; Glucocorticoids; Glucocorticoids Toxicity; Intravenous; Side effects; Adverse effects; Aminotransferase
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Liver Diseases; Liver Failure; Hepatic Insufficiency; Liver Failure, Acute; Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate-to-severe Graves Orbitopathy (Active Comparator): active, moderate-to-severe Graves Orbitopathy according to EUGOGO.
  Interventions: Drug: every week IVMP therapy
- Dysthyroid Orbit Neuropathy (Active Comparator): Dysthyroid Orbit Neuropathy according to EUGOGO
  Interventions: Drug: very high doses IVMP therapy

INTERVENTIONS:
Drug: every week IVMP therapy — 12 pulses of intravenous methylprednisolone (IVMP) in every week schedule (for the first 6 weeks 0.5g IVMP per week, for the next 6 weeks 0.25g IVMP per week; cumulative dose 4.5g) according to EUGOGO recommendations
  Arms: moderate-to-severe Graves Orbitopathy
Drug: very high doses IVMP therapy — 3 pulses of intravenous methylprednisolone (IVMP) (1.0g/day for 3 consecutive days; cumulative dose 3.0g) according to EUGOGO recommendations
  Arms: Dysthyroid Orbit Neuropathy

SUMMARY:
Graves' orbitopathy (GO) is a characterized by orbital soft tissue inflammation and oedema associated with glycosaminoglycan deposition and fibrosis. The most frequent cause is Graves' disease. The classification is comprised based on the severity of orbital changes ranging from mild, moderate-to-severe GO and sight-threatening GO, which includes dysthyroid optic neuropathy (DON). Intravenous methylprednisolone (IVMP) pulse therapy is the first-line treatment in the active-phase of moderate-to-severe GO and DON. This therapy is more effective and better tolerated than oral glucocorticoids (GCs). The current recommendation of the European Group of Graves' Orbitopathy (EUGOGO) is that cumulative doses of IVMP should not exceed 8.0g in each treatment course, and pulses should not be given on consecutive or alternate days, except in the case of DON. According to EUGOGO recommendations patients with moderate-to-severe GO are treated with IVMP cumulative dose 4.5g during a 12-week period (for the first 6 weeks 0.5g IVMP per week, for the next 6 weeks 0.25g IVMP per week). According to EUGOGO recommendations patients with DON should receive 3.0g IVMP (1.0g/day for 3 consecutive days) as the basic treatment. This limitation in doses are due to the necessity of the prevention of severe side effects that are rare but may be fatal. One of the most severe adverse events is acute liver injury (ALI), in some cases irreversible and/or fatal. The estimated morbidity and mortality of ALI was found to be 1-4 % and 0.01-0.3%, respectively. Since 2000, there were 5 reported fatal cases.

Mechanisms causing an IVMP-induced ALI remains incompletely elucidated. There are some possible hypotheses that may explain the occurrence of ALI. Firstly, GCs can lead to reactivation of autoimmune hepatitis: an immune "rebound phenomenon" following GCs withdrawal. The second mechanism of ALI is reactivation of viral hepatitis. Finally, there is well known direct toxic effect of GCs on hepatocytes, probably dose-dependent.

This study was performed to evaluate the influence of two different, routinely used schemes of therapy with IVMP in patients with moderate-to-severe GO (first scheme) and DON (second scheme) on biochemical liver parameters. Patients included into the study were treated according to EUGOGO recommendations with routine doses of IVMP and routine scheme of administration for moderate-to-severe GO and DON. No additional treatment was performed during the study protocol.

DETAILED DESCRIPTION:
Depending on the severity according to EUGOGO recommendations, patients were divided into two groups: the first group with active, moderate-to-severe GO (49 patients) and the second group with DON (19 patients). Moderate-to-severe GO was diagnosed according to EUGOGO recommendations. Diagnosis of DON in patients with GO was based on at least two signs, including (i) deterioration of VA (< 1.0), (ii) loss of colour vision (more than two errors in Ishihara plates), (iii) optic disc swelling, and/or (iv) signs of DON in a magnetic resonance (MR) scan (presence of apical crowding and/or optic nerve stretching).

Laboratory tests were performed before treatment in all patients from both evaluated groups. Serum markers of exposure to hepatitis B (HBV) and hepatitis C (HCV) were checked: hepatitis B surface antigen (HBs-Ag), hepatitis B surface antibody (HBs-Ab), hepatitis B core antibody (HBc-Ab), hepatitis C antibody (HCV-Ab). Serum autoantibodies associated with autoimmune hepatitis including anti-nuclear antibodies (ANA1), anti-smooth muscle antibodies (ASMA), anti-mitochondrial antibodies (AMA) and anti-liver kidney-microsomal antibodies (anti-LKM) were also assessed. Thyroid evaluation included measurement of: thyroid-stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), and serum antithyroid autoantibodies including anti-thyroid peroxidase (aTPO), thyroglobulin antibodies (aTG), thyroid-binding inhibitory immunoglobulin (TBII).

According to EUGOGO recommendations: patients with moderate-to-severe GO were treated with IVMP cumulative dose 4.5g during a 12-week period (for the first 6 weeks 0.5g IVMP per week was administrated and for the next 6 weeks 0.25g IVMP per week) and patients with DON received 3.0g IVMP (1.0g/day for 3 consecutive days).

Liver function parameters for further analysis included alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin. These parameters were measured the day before treatment in both groups and the day after administration of IVMP in selected pulses: after 0.5g (1st pulse), after 3.0g (6th pulse) and after 4.5g (12th pulse ) in the group with moderate-to-severe GO; after 3.0g IVMP in the group with DON.

Depending on concentrations of ALT, liver dysfunction was divided into: mild (above the upper limit of normal but less than 100 U/L), moderate (100-300 U/L) and severe (>300 U/L). ALI was defined as an ALT concentration >300 U/L. However, the investigators also evaluated a 4-fold increase of ALT in comparison to the initial values.

Routine laboratory tests and clinical evaluation were performed before every single pulse. Laboratory tests consisted of: ALT, AST, C reactive protein (CRP). In cases of moderate and severe increase in ALT (more than 100U/L) therapy was stopped.

Follow-up was performed in all of the patients and it included evaluation of AST, ALT and total bilirubin between 1-3 months after completion of IVMP therapy.

ELIGIBILITY:
Inclusion Criteria:

* active, moderate-to-severe Graves' orbitopathy or dysthyroid orbit neuropathy
* euthyroidism

Exclusion Criteria:

* alanine aminotransferase and/or aspartate aminotransferase >2x upper limit of normal
* active viral hepatitis
* cirrhosis
* present or past medical history of autoimmune hepatitis
* previous glucocorticoids therapy within the last 6 months
* alcohol abuse
* active inflammation
* active neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Influence of IVMP pulses in 12 every week schedule on mean ALT | 12 weeks
  Administration of IVMP in 12 every week schedule: 6 weeks 0.5g IVMP per week plus 6 weeks 0.25g IVMP per week. Change of mean value of alanine aminotransferase (ALT) between baseline (before administration of IVMP) and the end of the therapy (after the last pulse of IVMP).
Influence of IVMP pulses in 3 consecutive days schedule on mean ALT | 3 days
  Administration of 3g IVMP (1g in 3 consecutive days). Change of mean value of ALT between baseline (before IVMP) and the end of the therapy (after the last pulse of IVMP).

SECONDARY OUTCOMES:
Influence of IVMP pulses in 12 every week schedule on prevalence of mild, moderate and severe liver dysfunction. | 12 weeks
  Administration of IVMP in 12 every week schedule: 6 weeks 0.5g IVMP per week plus 6 weeks 0.25g IVMP per week. Depending on concentrations of ALT, liver dysfunction was divided into: mild (above the upper limit of normal but less than 100 U/L), moderate (100-300 U/L) and severe (>300 U/L). ALI was defined as an ALT concentration >300 U/L. Prevalence of all types of liver dysfunction was count after IVMP treatment.
Influence of IVMP pulses in 3 consecutive days schedule on prevalence of mild, moderate and severe liver dysfunction. | 3 days
  Administration of 3g IVMP (1g in 3 consecutive days). Depending on concentrations of ALT, liver dysfunction was divided into: mild (above the upper limit of normal but less than 100 U/L), moderate (100-300 U/L) and severe (>300 U/L). ALI was defined as an ALT concentration >300 U/L. Prevalence of all types of liver dysfunction was count after IVMP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Miśkiewicz, MD, PhD, Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The collected data will be shared in a publication.
Time Frame: The results of the study will be published in 2018-2019

REFERENCES:
- [Derived] Miskiewicz P, Jankowska A, Brodzinska K, Milczarek-Banach J, Ambroziak U. Influence of Methylprednisolone Pulse Therapy on Liver Function in Patients with Graves' Orbitopathy. Int J Endocrinol. 2018 Oct 21;2018:1978590. doi: 10.1155/2018/1978590. eCollection 2018. PMID 30420883